CLINICAL TRIAL: NCT01413763
Title: A Double-blind, Randomized, Placebo-controlled, 2-way Crossover Study to Assess the Potential Effect of Topically Applied Imiquimod Cream on Atrial Ectopy in Patients With Actinic Keratosis
Brief Title: Potential Effect of Topical Imiquimod on Atrial Ectopy in Patients With Actinic Keratosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: GW01-1001
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis; Atrial ectopy
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imiquimod cream (Active Comparator)
  Interventions: Drug: Imiquimod cream 3.75%
- Placebo cream (Placebo Comparator)
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Imiquimod cream 3.75% — 3.75% cream, applied daily for 2 weeks
  Arms: Imiquimod cream
Drug: Placebo cream — placebo cream applied daily for 2 weeks
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to determine the potential effect of topically applied 3.75% imiquimod cream on atrial ectopy in actinic keratosis (AK) patients. The primary endpoint is the change in the 24-hour supraventricular premature beat count. The secondary endpoint is the change in 24-hour supraventricular premature couplet and run counts and atrial fibrillation (% time); change in 24-hour mean heart rate; change in 24-hour ventricular premature beat count, ventricular premature couplet and run counts.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, 2-way crossover study designed to assess the potential effect of topically applied 3.75% imiquimod cream on atrial ectopy in actinic keratosis (AK) patients. Candidates for study participation will begin screening procedures up to 28 days prior to enrollment. Qualified subjects shall be admitted to the CRU on Day -1 for baseline evaluations and will be randomized to one of two possible treatment sequences. Each subject will receive both the active 3.75% imiquimod cream and the matching placebo in a randomized crossover fashion with a 2-week washout in between each treatment. The application area is the entire face (exclusive of nares, vermilion, periocular areas and ears) or balding scalp. Atrial ectopy will be monitored for 24 hours at Baseline (Day -1; prior to the first dose of study medication), and at the conclusion of each 14-day treatment period using a continuous 12-lead digital Holter recorder.

Adverse events, concomitant medication use, study medication accountability, and subject compliance will be reviewed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female AK patients with at least 5 typical visible or palpable AK lesions on face or balding scalp
* AK patients in otherwise good general health age 18 years and above
* Female subjects of childbearing potential must be non-pregnant and non-lactating

Exclusion Criteria:

* Previous clinical study participation within 30 days (drug or device)
* Evidence of clinically significant diseases
* History of drug or alcohol abuse
* Subjects with uncontrolled systemic hypertension, NYHA heart failure classification Class > II, or a history of atrial fibrillation or atrial flutter
* Subjects using imiquimod or interferon within 30 days prior to the first dose of study medication
* Have known allergies to any excipient in the study cream
* Have melanoma anywhere on the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour supraventricular beat count | Day 14 of each treatment period

SECONDARY OUTCOMES:
Change in 24-hour supraventricular premature couplet and run counts and atrial fibrillation (% time) | Day 14 of each treatment period
Change in 24-hour mean heart rate | Day 14 of each treatment period
Change in 24-hour ventricular premature beat count, ventricular premature couplet and run counts | Day 14 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Babilon, MS, MBA, Study Director — Graceway Pharmaceuticals, LLC
Locations (1):
- Comprehensive Phase One, Fort Meyers, Florida, United States